CLINICAL TRIAL: NCT03985930
Title: Non-immersive Virtual Reality for Pediatric Pain Management
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Claudia Aristizábal (Other)
Collaborators: Sanitas University (Other)
Responsible Party: Sponsor-Investigator, Claudia Aristizábal, Coordinadora Unidad de Investigación, Sanitas University
Organization: Sanitas University (Other)
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: VRPedPain
Record Dates: First submitted 2019-06-11; First posted 2019-06-14 (Actual); Last update posted 2023-04-03 (Actual); Status verified 2023-03

CONDITIONS: Procedural Pain
Keywords: Child, Preschool; Virtual Reality; Procedural Pain; Phlebotomy; Vaccination
MeSH Terms: conditions — Pain, Procedural | interventions — Therapeutics

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Distraction Group (Experimental): Children between the ages of 3 and 5 years will be distracted using virtual reality content delivered through goggles.
  Interventions: Device: Distraction with virtual reality
- Treatment as Usual (Active Comparator): Children randomized to this group will receive the usual medical care.
  Interventions: Other: Treatment as Usual

INTERVENTIONS:
Device: Distraction with virtual reality — Distraction content delivered through virtual reality goggles
  Arms: Distraction Group
Other: Treatment as Usual — Treatment as Usual
  Arms: Treatment as Usual

SUMMARY:
This is a multicenter, randomized, clinical trial comparing treatment as usual to distraction with video projection or virtual reality in the management of pediatric (3-6 years) pain associated with venipuncture, intramuscular injection, and vaccination.

DETAILED DESCRIPTION:
Background: Recent studies have shown that the use of virtual reality (VR) may be useful to provide distraction that attenuates pain in minimally invasive procedures in preschool children.

Aim: To assess the effectiveness of non-immersive virtual reality as a pain-distraction measure in children between the ages of 3 to 5 years undergoing painful injection procedures in an outpatient setting.

Method: This clinical trial will recruit patients under 6 years of age treated at participating medical centers in whom a painful procedure like vaccination, venipuncture or administration of intramuscular medication will be performed. The experimental group will consist of two subgroups which, in addition to treatment as usual, will be distracted using virtual reality content delivered through goggles. The control group will receive treatment as usual. The LLANTO pain scale will be used to measure different characteristics of pain. This scale has been validated in Colombia, and will be filled by two health professionals (one of which will perform the painful procedure.) and the parents.

Expected results: To show that virtual reality or projector distraction are effective distraction tools in pain management for children subjected to painful procedures of venipuncture, intramuscular medication administration, and vaccination.

ELIGIBILITY:
Inclusion Criteria:

* Patients subjected to procedures of venipuncture, intramuscular injections, or vaccination at participating medical centers.

Exclusion Criteria:

* Fever (Axillary temperature greater than 38°C).
* Systemic Inflammatory Response Syndrome or Sepsis.
* Pulmonary disease.
* Neurological deficit of any kind.
* Susspected or confirmed metabolic disease.
* Undernutrition or obesity as defined by deviations from the mean of local values.

Ages: 3 Years to 5 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Enrollment: 122 (Actual)
Dates: Start 2020-11-01 (Actual); Primary Completion 2021-11-01 (Actual); Study Completion 2021-12-01 (Actual)

PRIMARY OUTCOMES:
LLANTO Pain level: LLANTO pain scale | Immediately after procedure
  Overall pain assessment using the LLANTO pain scale (Mild: 0-3, Moderate 4-6, Intense 7-10) For more information about LLANTO scale, please visit DOI: 10.1016/j.anpedi.2010.08.005

SECONDARY OUTCOMES:
LLANTO Crying | Immediately after procedure
  Subcomponent of the LLANTO scale scored as not crying (0), crying but consolable (1), or insconsolable crying (2).
LLANTO Attitude | Immediately after procedure
  Subcomponent of the LLANTO scale scored as at ease or sleeping (0), restless (1), or agressive (2).
LLANTO Breathing | Immediately after procedure
  Subcomponent of the LLANTO scale scored normal (0), tachypneic (1), or irregular (2).
LLANTO Facial expression | Immediately after procedure
  Subcomponent of the LLANTO scale scored content or sleeping (0), unsmiling (1), or unhappy (2).
LLANTO Postural muscle tone | Immediately after procedure
  Subcomponent of the LLANTO scale scored as relaxed (0), indifferent (1), or contracted (2).
Interrater reliability of the LLANTO scale | During the statistical analysis stage
  Between parents, nurse and physician

CONTACTS AND LOCATIONS:
Overall Officials: Jhon H Camacho Cruz, M.D., Principal Investigator — Fundación Universitaria Sanitas
Locations (1):
- Fundación Universitaria Sanitas, Bogotá, Bogota D.C., Colombia

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Camacho-Cruz J, Palacios-Ariza MA, Orrego-Celestino L, Valbuena-Velandia N, Paez-Castellanos L, Bolanos JM, Pradilla I. Effectiveness of non-immersive virtual reality in the management of procedure-related pain in preschool children: a randomized clinical trial. Eur J Pediatr. 2023 Sep;182(9):4103-4112. doi: 10.1007/s00431-023-05070-5. Epub 2023 Jul 5. PMID 37407711